CLINICAL TRIAL: NCT04474847
Title: A Randomized Double-Blind, Placebo Controlled Trial of Abatacept (CTLA4-Ig) in Giant Cell Arteritis (ABAGART)
Brief Title: Abatacept for the Treatment of Giant Cell Arteritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCRC5528
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Giant Cell Arteritis
Keywords: Vasculitis; Arteritis; Temporal Arteritis; Abatacept; CTLA4-Ig; Autoimmune Diseases; Immune System Diseases; Immunosuppressive agent; Prednisone; Glucocorticoids; Corticosteroids; Treatment; Pharmacologic Actions; Therapeutic Uses; Anti Inflammatory Agents; Antirheumatic Agents
MeSH Terms: conditions — Giant Cell Arteritis; Vasculitis; Arteritis; Autoimmune Diseases; Immune System Diseases | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Blinded Abatacept (Experimental): Participants will receive blinded abatacept 125 mg administered by subcutaneous injection once a week for at least 12 months. Subjects may be removed from treatment earlier due to a disease relapse, disease worsening, or if they have not achieved remission.
  Interventions: Drug: Abatacept
- Blinded Placebo (Placebo Comparator): Participants will receive blinded placebo. Placebo will be administered by subcutaneous injection once a week for at least 12 months. Subjects may be removed from treatment earlier due to a disease relapse, disease worsening, or if they have not achieved remission.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept — Participants randomized to abatacept will receive abatacept 125 mg administered by subcutaneous injection once a week. Participants randomized to either the abatacept or the placebo arm who experience a non-severe disease relapse, non-severe disease worsening, or who have not achieved remission by month 3 will have the option of entering an open-label trial period whereby they would receive open-label abatacept for up to 12 months.
  Other Names: CTLA4-Ig; Orencia
  Arms: Blinded Abatacept
Drug: Placebo — Participants randomized to placebo will receive a sterile placebo solution administered by subcutaneous injection once a week. Participants randomized to either the abatacept or the placebo arm who experience a non-severe disease relapse, non-severe disease worsening, or who have not achieved remission by month 3 will have the option of entering an open-label trial period whereby they would receive open-label abatacept for up to 12 months.
  Arms: Blinded Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled trial will seek to determine the efficacy of abatacept in GCA. To examine this objective, 62 eligible patients who have newly diagnosed or relapsing GCA within 8 weeks prior to screening will be randomized at a 1:1 ratio to receive subcutaneous abatacept 125mg/week or placebo. Patients who achieve remission will remain on their blinded assignment for 12 months at which time abatacept/placebo will be stopped.

Patients who do not achieve remission by Month 3, who experience a relapse within the first 12 months will have the option of receiving open-label abatacept for a maximum of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of newly diagnosed or relapsing GCA. Diagnostic criteria for GCA

   A patient will be said to have GCA by meeting 3 of 5 of the following modified ACR criteria for the classification of GCA in which 1 of the 3 must consist of criteria 4 or 5:
   1. Age at disease onset ≥ 50 years.
   2. New onset or new type of localized pain in the head.
   3. ESR of > 40 mm in the first hour by the Westergren method or CRP measurement above the laboratory normal limit.
   4. Temporal artery abnormality (i.e., temporal artery tenderness to palpation or decreased pulsation, unrelated to arteriosclerosis of cervical arteries).
   5. Temporal artery or large vessel biopsy showing vasculitis characterized by a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cell or an abnormal temporal artery ultrasound showing features consistent with active giant cell arteritis ("halo sign") or characteristic changes of large vessel stenosis or aneurysm by arteriography.
2. GCA with evidence of active disease (defined below) present within the past 8 weeks.
3. They must be willing and able to comply with treatment and follow-up procedures.
4. Both women and men who are of child-bearing potential must be willing to use an effective means of birth control while receiving treatment through this study. Effective contraception methods include abstinence, surgical sterilization of either partner, barrier methods such as diaphragm, condom, cap or sponge, or hormonal contraception.
5. They must be willing and able to provide written informed consent.

Exclusion Criteria:

1. Evidence of a recent acute infection defined as:

   * Any acute infection within 60 days prior to randomization that required hospitalization or treatment with parenteral antibiotics.
   * Any acute infection within 30 days prior to randomization that required oral antimicrobial or antiviral therapy.
2. Patients with history of chronic or recurrent bacterial infection (such as chronic pyelonephritis, osteomyelitis, and bronchiectasis etc.).
3. Patients with a history of recurrent herpes zoster (more than 1 episode) or disseminated (more than 1 dermatome) herpes zoster or disseminated herpes simplex, or ophthalmic zoster. Symptoms of herpes zoster or herpes simplex must have resolved more than 60 days prior to screening.
4. Patients with a history of systemic fungal infections (such as histoplasmosis, blastomycosis, or coccidiomycosis).
5. Patients with a history of primary immunodeficiency.
6. Patients at risk for tuberculosis (TB) defined as follows:

   * Current clinical, radiographic or laboratory evidence of active TB, even if currently being treated. Chest x-rays (posterior/anterior and lateral) obtained within the 6 months prior to screening and TB testing (IFN-gamma release assay or PPD) performed in the past month prior to screening will be accepted; however, a copy of the reports must be placed in the participant binder.
   * A history of active TB unless there is documentation that the patient had received prior anti-TB treatment that was appropriate in duration and type according to local health authority guidelines.
   * Patients with a positive TB screening test indicative of latent TB will not be eligible for the study unless they:

     i. Have no evidence of current TB based on chest x-ray performed during the screening period and by history and physical exam, and ii. They are currently being treated for latent TB or the site has documentation of successful prior treatment of latent TB. Treatment regimens should be dictated by local guidelines as long as the treatment dose and duration meet or exceed local health authority guidelines. If permitted by local guidelines regarding treatment with biologic medications, patients with latent TB may be randomized prior to completion of treatment as long as they have completed at least 4 weeks of treatment and they have no evidence of current TB on chest x-ray at screening.
7. Patients who are pregnant or who are nursing infants.
8. Inability to comply with study guidelines.
9. Cytopenia: platelet count <80,000/mm3, total White Blood Count (WBC) < 3,000/mm3 (3 x 109/L) absolute neutrophil <1500/mm3, hematocrit < 20%.
10. Renal insufficiency defined by a creatinine clearance of less than or equal to 20 ml/min.
11. AST or ALT > 3 times above normal laboratory range.
12. Other severe, progressive, or uncontrolled disease that in the investigator's opinion could prevent a patient from fulfilling the study requirements or that would increase the risk of study participation.
13. Patients who have a present malignancy or previous malignancy within the last 5 years prior to screening (except documented history of cured non-metastatic squamous or basal cell skin carcinoma or cervical carcinoma in situ). Patients who had a screening procedure that is suspicious for malignancy, and in whom the possibility of malignancy cannot be reasonably excluded following additional clinical, laboratory or other diagnostic evaluations.
14. Receipt of an investigational agent or device within 30 days prior to enrollment.
15. A live vaccination within 3 months before randomization.
16. Patients on non-biologic immunosuppressants must discontinue these medications before randomization (azathioprine, mycophenolate mofetil, mycophenolic acid, leflunomide, hydroxychloroquine, cyclosporin, tacrolimus, or other conventional immunosuppressive agent).
17. Patients who had received an alkylating agent such as cyclophosphamide must discontinue these medications at least 8 weeks before randomization.
18. Patients who have been treated within 4 weeks of randomization with etanercept or within 8 weeks with adalimumab, certolizumab, golimumab, or infliximab.
19. Patients who have been treated within 8 weeks of randomization with anti-IL-6 agents (e.g., tocilizumab, sirukumab) or a janus kinase inhibitor.
20. Patients who have been treated within 4 weeks of randomization with anakinra.
21. Patients who have received prior treatment with rituximab within the past 6 months prior to randomization.
22. Patients who have received prior treatment with abatacept or CTLA4-Ig.
23. Patients who will require oral or IV glucocorticoid treatment during the trial for conditions other than GCA.
24. Hypersensitivity to abatacept and/or its excipients.
25. Presence of any of the following disease processes:

    * Takayasu arteritis
    * Granulomatosis with polyangiitis
    * Microscopic polyangiitis
    * Eosinophilic granulomatosis with polyangiitis (Churg-Strauss)
    * Polyarteritis nodosa
    * Cogan's syndrome
    * Behçet's disease
    * Sarcoidosis
    * Lymphoma, lymphomatoid granulomatosis, or other type of malignancy that mimics vasculitis
    * Cryoglobulinemic vasculitis
    * Systemic lupus erythematosus
    * Rheumatoid arthritis
    * Mixed connective tissue disease or any overlap autoimmune syndrome

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants in remission of those randomized to abatacept as compared to placebo. | 12 months
  Remission is defined as the absence of clinical or imaging features of active disease

SECONDARY OUTCOMES:
Safety of abatacept in GCA | 12 months
  Safety of abatacept in patients with GCA as assessed by reported adverse events.
Health-related quality of life in those treated with abatacept versus placebo: SF-36 | 12 months
  Health-related quality of life in those treated with abatacept versus placebo as assessed using the SF-36
Health-related quality of life in those treated with abatacept versus placebo: PROMIS questionnaire | 12 months
  Health-related quality of life in those treated with abatacept versus placebo as assessed using a PROMIS questionnaire
Duration of glucocorticoid-free remission from Month 6 to Month 12 | 6 months
  Effect of abatacept on increasing duration of glucocorticoid-free periods for participants.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Merkel, MD, MPH, Principal Investigator — University of Pennsylvania; Carol A Langford, MD, MHS, Principal Investigator — The Cleveland Clinic; Jeffrey P Krischer, PhD, Principal Investigator — University of South Florida
Locations (9):
- United States (5):
  - Mayo Clinic, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hôpital du Sacré-Coeur de Montréal Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No